CLINICAL TRIAL: NCT00003732
Title: A Phase I/II Study to Determine the Maximum Tolerated Doses of Oral Topotecan, Carboplatin and Paclitaxel Administered Every 21 Days to Patients With Epithelial Ovarian Cancer Stages IIb, IIc, III and IV
Brief Title: Combination Chemotherapy in Treating Patients With Stage II, Stage III, or Stage IV Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DAN-104864/373; CDR0000066847 (Registry Identifier: PDQ (Physician Data Query)); DAN-104864-A/373; EU-98052; SB-104864-A/373; SB-104864/373
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2002-07

CONDITIONS: Ovarian Cancer
Keywords: stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel; Topotecan

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of topotecan combined with carboplatin and paclitaxel in treating patients who have stage II, stage III, or stage IV ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, dose-limiting toxicity, and quantitative and qualitative toxic effects of oral topotecan combined with intravenous carboplatin and paclitaxel in patients with stage IIB, IIC, III, or IV ovarian epithelial cancer. (phase I closed to accrual 12/21/00)
* Evaluate the anti-tumor activity of this regimen in this patient population.

OUTLINE: This is a multicenter, dose-escalation study of topotecan.

Patients receive oral topotecan on days 1-5 and paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 5. Courses repeat every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

* Phase I: Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. (phase I closed to accrual 12/21/00)
* Phase II: An additional 50 patients receive up to 6 courses of treatment as in phase I at the MTD.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 80 patients (30 in phase I and 50 in phase II) will be accrued for this study. (phase I closed to accrual 12/21/00)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIB, IIC, III, or IV ovarian epithelial cancer
* Measurable or evaluable lesion or microscopic residual disease after first surgery (phase II patients)
* No brain and/or leptomeningeal metastases by CT scan or MRI unless asymptomatic without corticosteroid therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 9.0 g/dL
* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) unless liver metastases present
* Alkaline phosphatase no greater than 2 times ULN*
* SGOT no greater than 2 times ULN* NOTE: *No greater than 5 times ULN if liver metastases present

Renal:

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic cardiac disease, including clinical congestive heart failure or arrhythmias requiring treatment
* No myocardial infarction within the past 3 months

Other:

* No other malignancy except basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled infection
* No complete bowel obstruction or other condition that would affect GI absorption or motility
* No concurrent medical condition for which treatment with platinum, taxane, or camptothecin analogues are contraindicated
* No other concurrent medical conditions that would preclude study
* No mental disease
* No history of allergy to platinum or taxanes, including drugs containing cremophor (e.g., cyclosporine or vitamin K)
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior camptothecin analogue
* No prior chemotherapy for ovarian cancer
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent hormonal therapy other than estrogen replacement

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 30 days or 5 half-lives since any prior investigational therapy
* No other concurrent investigational therapy
* No concurrent metoclopramide or cisapride

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1998-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of topotecan
Toxic effects
Antitumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Svend Aage Engelholm, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark